CLINICAL TRIAL: NCT06713629
Title: The Use of PlCO-Vacuum-System on Sternal Wounds
Acronym: PICO sternal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Smith & Nephew, Inc. (Industry); Kerckhoff Heart Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ 62/19
Record Dates: First submitted 2024-04-09; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgery; Wound Infection; Wound Healing Disorder
Keywords: vacuum wound dressing; PICO; sternal wound healing disorder
MeSH Terms: conditions — Wound Infection | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICO arm (Experimental): PICO vacuum system for post-sternotomy wound
  Interventions: Procedure: cardiac surgery via median sternotomy
- Control arm (Active Comparator): usual commercial wound dressing
  Interventions: Procedure: cardiac surgery via median sternotomy

INTERVENTIONS:
Procedure: cardiac surgery via median sternotomy — For both groups, the same median sternotomy cardiac surgery procedure
  Other Names: wound dressing; PlCO-Vacuum dressing

SUMMARY:
The use of a vacuum-assisted wound closure system (PICO, Fa. Smith & Nephew) is being investigated to determine whether it reduces the incidence of sternal wound healing disorders compared to conventional wound care with plaster.

DETAILED DESCRIPTION:
Median sternotomy remains the standard surgical approach for most cardiac surgeries. However, postoperative wound infections can occur and may progress to mediastinitis, a life-threatening complication with significant mortality. This risk is particularly pronounced in cases where sternal perfusion is compromised, such as when one or both internal mammary arteries are harvested during coronary artery bypass grafting. In such scenarios, the incidence of sternal wound healing disturbances is estimated to range from 2% to 7%.

Several strategies aim to reduce the risk of sternal wound infections. One approach involves external stabilization using a thoracic vest, which has been shown to significantly decrease sternal instability and healing disorders when implemented early in the postoperative period. Another approach utilizes negative pressure wound therapy, which has demonstrated efficacy in reducing sternal wound healing complications in prior studies involving systems like Prevena (Fa. KCI).

The PICO-System operates with a distinct vacuum pressure mechanism and a unique film design compared to the Prevena system. To date, no prospective randomized studies have evaluated the PICO-System for its effectiveness in reducing sternal healing disturbances, sternal instability, and mediastinitis. This study aims to compare conventional plaster wound care with the PICO vacuum system in a randomized, prospective design, assessing outcomes up to six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing cardiac surgery by means of median sternotomy and exhibiting more than one of the following risk factors:

* Diabetes mellitus (treated with oral antidiabetics and/or insulin)
* LVEF<40%
* COPD
* Female gender
* Adipositas (BMI > 30kg/m2)
* History of myocardial infarction (NSTEMI or STEMI) within 14 days
* Known peripheral arterial disease
* Planned BIMA surgery.

Exclusion Criteria:

* Planned hemisternotomy or anterolateral thoracotomy
* Emergency cases
* Lack of consent
* Active therapy with immunosuppressants (including steroids)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Infection at 30 POD | until day 30 post-surgery
  Rate of superficial or deep sternal wound healing disorders at 30 days postoperatively

SECONDARY OUTCOMES:
Infection at 180 Postoperative Days (POD) | Up to 180 days post-surgery
  Rates of superficial and/or deep sternal wound healing disorders assessed using standardized clinical criteria, including infection signs (e.g., erythema, purulent discharge), radiological imaging (if indicated), microbiological culture results, and adherence to validated classification systems such as the CDC's surgical site infection (SSI) criteria.
Patient satisfaction | until day 7 post-surgery
  Patient satisfaction with the PICO-System in comparison to conventional plasters:
  The following questions were assessed to evaluate participant satisfaction:
  * The wound dressing causes discomfort.
  * My wound has achieved a satisfactory cosmetic appearance.
  * I experienced pain during wound dressing changes.
  * I am generally satisfied with the care provided.
  For each question, the following response options were offered:
  * Fully applies
  * Partially applies
  * Neutral
  * Partially does not apply
  * Does not apply

OTHER OUTCOMES:
Cost-Effectiveness of PICO Wound Dressing Compared to Conventional Plaster Dressing | From surgery to day 180 post-surgery
  The cost-effectiveness analysis will assess the direct and indirect costs associated with the use of PICO vacuum-assisted wound dressings compared to conventional plaster dressings in patients undergoing median sternotomy. Costs will include initial purchase price, frequency of dressing changes, associated resource utilization (e.g., hospital readmissions, additional interventions for wound healing disorders), and postoperative complications such as sternal instability, wound infections, and mediastinitis. Data will be aggregated and reported using descriptive statistics, incremental cost-effectiveness ratios.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Cardiac Surgery, Kerckhoff Heart Center, Bad Nauheim, Hesse
  - Cardiovascular Surgery, University Hospital Giessen, Giessen, Hesse

IPD SHARING:
Plan to Share IPD: No